CLINICAL TRIAL: NCT00410410
Title: A Phase 3, Multi-Center, Randomized, Placebo-Controlled Study to Evaluate the Clinical Efficacy and Safety of Induction and Maintenance Therapy With Abatacept in Subjects With Active Ulcerative Colitis (UC) Who Have Had an Inadequate Clinical Response and/or Intolerance to Medical Therapy
Brief Title: A Study of Abatacept in Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-108
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Abatacept (ABA) (Experimental): Induction Period; 3 arms for Cohort 1: ABA 30/~10 mg/kg (ABA administered at 30 mg/kg followed by ABA at ~10 mg/kg), ABA ~10 mg/kg, ABA 3 mg/kg
  Induction Period; 2 arms for Cohort 2: ABA 30/~10 mg/kg and Second Cohort ABA ~10 mg/kg
  1 arm for maintenance period (ABA ~10 mg/kg)
  Interventions: Drug: abatacept (ABA)
- Placebo (Placebo Comparator): 1 arm for induction period
  1 arm for maintenance period
  Interventions: Drug: placebo
- abatacept (Other): 1 arm for open-label extension phase (ABA ~10 mg/kg)
  Interventions: Drug: abatacept

INTERVENTIONS:
Drug: abatacept (ABA) — Dextrose 5% in water, IV. Placebo on days IP-1, IP-15,IP-29, IP-57; 3 mg/kg on days IP-1, IP-15,IP-29, IP-57; 10 mg/kg on days IP-1, IP-15,IP-29, IP-57; or 30 mg/kg on days IP-1,IP-15 and ~10 mg/kg on days IP-29, IP-57 (ABA 30/~10 mg/kg Group).
  Induction Period 3 months
  Maintenance Period 12 months
  Other Names: Orencia; BMS-188667
  Arms: Abatacept (ABA)
Drug: placebo — Normal saline, IV, 0 mg/kg, every 28 days.
  Induction Period 3 months
  Maintenance Period 12 months
  Arms: Placebo
Drug: abatacept — ~10 mg/kg, once monthly
  Open- Label Extension Period until the drug is marketed for UC or the UC development program for abatacept is discontinued
  Other Names: Orencia; BMS-188667
  Arms: abatacept

SUMMARY:
The purpose of this clinical research study is to learn if abatacept can improve signs and symptoms of active ulcerative colitis in patients who have not had an adequate response to other therapies. The safety of this treatment will also be studied

DETAILED DESCRIPTION:
The Induction Period First Cohort (IP1C) arms (30/10 mg/kg and 10 mg/kg) were placebo-controlled arms that were used for the primary endpoint and its analysis. The Induction Period Second Cohort arms (IP2C 30/10 mg/kg and 10 mg/kg) were not placebo-controlled, their sole purpose being to provide sufficient numbers of participants for the maintenance phase. The first cohort (IP1C) was randomized to receive placebo or 1 of 3 doses of abatacept. Following completion of the IP1C randomization, a second cohort (IP2C) was randomized to receive 1 of 2 doses of abatacept. After all participants in the IP1C completed or discontinued, the data was locked and the formal analysis for the Induction Period primary endpoint was performed. Summary tables for the second cohort (IP2C) and the Maintenance and Open-label phases were generated from a second, subsequent data lock.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years or older
* Ulcerative colitis for at lease 3 months
* Moderate to severe active ulcerative colitis
* Inadequate response or intolerance to standard ulcerative colitis treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (131):
- United States (50):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Permanente Medical Group, Inc, Sacramento, California
  - Western States Clinical Research Inc., Wheat Ridge, Colorado
  - Litchfield County Gastroenterology Assoc., Torrington, Connecticut
  - University Of Florida, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - Shafran Gasteroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University Of Chicago Hospitals, Chicago, Illinois
  - Health Science Center, Pratt, Kansas
  - University Of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Gulf Coast Research, Lafayette, Louisiana
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Kansas City Gastroenterology And Hepatology, Kansas City, Missouri
  - Center For Digestive & Liver Diseases, Inc., Mexico, Missouri
  - Aga Clinical Research Associates, Llc, Egg Harbor Twp, New Jersey
  - Hudson Valley Medical Research Llc, Fishkill, New York
  - Long Island Clinical Research, Great Neck, New York
  - Mount Sinai School Of Medicine, New York, New York
  - University Of Rochester Medical Center, Rochester, New York
  - Good, Larry I., Rockville Centre, New York
  - Gastrointestinal Resrch Assoc., Setauket, New York
  - University Of North Carolina, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, Pllc, Charlotte, North Carolina
  - Hanover Medical Specialists, P.A., Wilmington, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Gastroenterology Specialists, Inc., Canton, Ohio
  - Consultants For Clinical Research, Inc., Cincinnati, Ohio
  - Gastrointestinal & Liver Diseases Consultants, Dayton, Ohio
  - Oklahoma Foundation For Digestive Research, Oklahoma City, Oklahoma
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Center For Digestive Health, Pittsburgh, Pennsylvania
  - Medical University Of South Carolina, Charleston, South Carolina
  - Gastroenterology Center Of The Midsouth, P.C., Germantown, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Nashville Medical Research, Nashville, Tennessee
  - Austin Gastroenterology, Pa, Austin, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Gastroenterology Clinic Of San Antonio, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Tacoma Digestive Disease Research Ctr., Tacoma, Washington
- Australia (10):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Herston, Queensland
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Launceston, Tasmania
  - Local Institution, Box Hill, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, South Ballarat, Victoria
  - Local Institution, Fremantle, Western Australia
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- Brazil (9):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Goiânia, Goiás
  - Local Institution, Curitiba, Paraná
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, Santo Andre - Sp, São Paulo
  - Local Institution, Santos, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (8):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Kingston, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Lévis, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Czechia (2):
  - Local Institution, Brno-Bohunice
  - Local Institution, České Budějovice
- France (7):
  - Local Institution, Amiens
  - Local Institution, Clichy
  - Local Institution, Lille
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Toulouse
- Germany (2):
  - Local Institution, Kiel
  - Local Institution, Münster
- India (10):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Kochi, Kerala
  - Local Institution, Mumbai, Maharashtra
  - Local Institution, Bangalore
  - Local Institution, Delhi
  - Local Institution, Hyderabad
  - Local Institution, Mangalore
  - Local Institution, Manipal
  - Local Institution, Mumbai
  - Local Institution, Mysore
- Local Institution, Dublin, Dublin, Ireland
- Italy (4):
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, San Giovanni Rotondo
- Mexico (9):
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Torreón, Coahuila
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Mexico, D. F., Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Hermosillo, Sonora
- Netherlands (3):
  - Local Institution, Amersfoort
  - Local Institution, Amsterdam
  - Local Institution, Groningen
- Poland (3):
  - Local Institution, Katowice
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Local Institution, Ponce, Puerto Rico
- South Africa (5):
  - Local Institution, Parktown West, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Overport, KwaZulu-Natal
  - Local Institution, Belville, Western Cape
  - Local Institution, Panorama, Western Cape
- Local Institution, Seoul, South Korea
- Switzerland (2):
  - Local Institution, Bern
  - Local Institution, Zurich
- United Kingdom (2):
  - Local Institution, London, Greater London
  - Local Institution, Oxford, Oxfordshire

REFERENCES:
- [Derived] Sandborn WJ, Colombel JF, Sands BE, Rutgeerts P, Targan SR, Panaccione R, Bressler B, Geboes K, Schreiber S, Aranda R, Gujrathi S, Luo A, Peng Y, Salter-Cid L, Hanauer SB. Abatacept for Crohn's disease and ulcerative colitis. Gastroenterology. 2012 Jul;143(1):62-69.e4. doi: 10.1053/j.gastro.2012.04.010. Epub 2012 Apr 12. PMID 22504093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, a first cohort (Induction Period First Cohort, IP1C) of 490 participants was randomized and used for analysis of the primary endpoint. Following randomization of IP1C, a second cohort (IP2C) of 146 participants was randomized to provide a sufficient number of participants for the Maintenance Period.
Groups:
- Induction Period Cohort 1 (IP1C)-Abatacept (ABA) 30/~10 mg/kg; IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). Following this, on Days IP-29 and IP-57 abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
- IP1C-ABA ~10 mg/kg; IP2C-ABA ~10 mg/kg: During IP, abatacept was administered IV on Days IP-1,IP-15, IP-29, and IP-57 at a dose of ~10 mg/kg (weight-tiered).
- IP1C-ABA 3 mg/kg: During IP, abatacept was administered IV on Days IP-1, IP-15, IP-29, and IP-57 at a dose of 3 mg/kg (fixed dose).
- IP1C-Placebo: During the IP, placebo was administered IV on Days IP-1, IP-15, IP-29, and IP-57.
- ABA ~10 mg/kg, Maintenance Period (MP): During MP, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered) every 28 days beginning Day MP-1.
- Placebo, MP: During the MP, placebo was administered IV every 28 days beginning Day MP-1 through Day MP-337.
- ABA ~10 mg/kg, Open-Label Period (OL): During OL, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered) every 28 days beginning Day OL-1.
Period: Induction Period (IP)
Arm/Group | Induction Period Cohort 1 (IP1C)-Abatacept (ABA) 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo | IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg | ABA ~10 mg/kg, Maintenance Period (MP) | Placebo, MP | ABA ~10 mg/kg, Open-Label Period (OL)
Started | 141 | 139 | 70 | 140 | 51 | 50 | 0 | 0 | 0
Completed | 106 | 104 | 53 | 120 | 19 | 21 | 0 | 0 | 0
Not Completed | 35 | 35 | 17 | 20 | 32 | 29 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 4 | 2 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 26 | 24 | 8 | 8 | 7 | 7 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 2 | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 3 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Subject No Longer Meets Study Criteria | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative Reason By Sponsor | 0 | 0 | 0 | 0 | 22 | 21 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (MP)
Arm/Group | Induction Period Cohort 1 (IP1C)-Abatacept (ABA) 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo | IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg | ABA ~10 mg/kg, Maintenance Period (MP) | Placebo, MP | ABA ~10 mg/kg, Open-Label Period (OL)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 65 (At end of IP, 65 participants met response criteria and were randomly assigned to abatacept in MP.) | 66 (At end of IP, 66 participants met response criteria and were randomly assigned to placebo in MP.) | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 11 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 55 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 24 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Administrative Reason By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 25 | 0
Period: Open-Label Period (OL)
Arm/Group | Induction Period Cohort 1 (IP1C)-Abatacept (ABA) 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo | IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg | ABA ~10 mg/kg, Maintenance Period (MP) | Placebo, MP | ABA ~10 mg/kg, Open-Label Period (OL)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 349 (349 entered OL (those who completed IP but failed response criteria, or completed/relapsed on MP).)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 349
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 161
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Administrative Reason By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 145
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg; IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). Following this, on Days IP-29 and IP-57 abatacept was administered IV at a dose of ~10 mg/kg.
- IP1C-ABA ~10 mg/kg; IP2C-ABA ~10 mg/kg: During IP, abatacept was administered IV on Days IP-1,IP-15, IP-29,and IP-57 at a dose of ~10 mg/kg (weight-tiered).
- Total: Total of all reporting groups
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo | IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg | Total
Number analyzed (Participants) | 141 | 139 | 70 | 140 | 51 | 50 | 591
Age, Customized [Number; unit: participants]
  <30 years | 26 | 23 | 18 | 34 | 12 | 4 | 117
  30-50 years | 70 | 84 | 35 | 73 | 30 | 32 | 324
  >50 years | 45 | 32 | 17 | 33 | 9 | 14 | 150
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 52 | 26 | 66 | 21 | 26 | 248
  Male | 84 | 87 | 44 | 74 | 30 | 24 | 343
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 22 | 55 | 20 | 13 | 195
  Ireland | 1 | 0 | 0 | 1 | 0 | 1 | 3
  Italy | 7 | 6 | 2 | 3 | 2 | 1 | 21
  Switzerland | 1 | 1 | 1 | 2 | 1 | 0 | 6
  United Kingdom | 0 | 0 | 0 | 3 | 2 | 4 | 9
  India | 12 | 12 | 10 | 10 | 5 | 2 | 51
  France | 7 | 12 | 6 | 6 | 1 | 5 | 37
  Czech Republic | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Mexico | 20 | 14 | 10 | 8 | 7 | 9 | 68
  Puerto Rico | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Canada | 9 | 12 | 2 | 13 | 1 | 3 | 40
  Brazil | 10 | 5 | 5 | 11 | 4 | 6 | 41
  Poland | 2 | 2 | 0 | 1 | 1 | 0 | 6
  Belgium | 4 | 6 | 1 | 5 | 0 | 1 | 17
  Australia | 8 | 7 | 4 | 13 | 1 | 1 | 34
  South Africa | 9 | 8 | 5 | 3 | 2 | 0 | 27
  Germany | 2 | 2 | 0 | 1 | 2 | 2 | 9
  Netherlands | 2 | 5 | 1 | 2 | 2 | 1 | 13
  Korea, Republic of | 4 | 3 | 1 | 2 | 0 | 1 | 11
Participants with Inadequate Response/Intolerance to Prior Anti-Tumor (TNF) Therapy (Infliximab) [Number; unit: participants] — Prior to this study, participants had an inadequate response and/or intolerance to an approved anti-TNF agent at an approved labeled dose for at least 8 weeks. Inadequate response was assessed by the treating physician and was primarily due to lack of efficacy. Because the treating physician determined prior inadequate response, there was no standard definition for this and criteria for determination may have varied between institutions. Intolerance was defined a an inability to achieve doses or treatment durations because of dose limiting side effects.
  participants
    Inadequate Response/Intolerant to prior Infliximab | 45 | 46 | 24 | 45 | 21 | 21 | 202
    No Inadequate Response/Intolerance to Infliximab | 96 | 93 | 46 | 95 | 30 | 29 | 389

OUTCOME MEASURES:

1. Primary Outcome: Induction Period (IP); Number of Participants With Clinical Response (Per Mayo Score) at Week 12: IP Cohort 1 (IP1C)
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. A clinical response is defined as a reduction from baseline in the Mayo score of ≥ 3 points and ≥ 30%, with an accompanying decrease in the rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point.
Time Frame: Week 12 (Day IP-85)
Population: All participants who were randomized and received at least one infusion of study medication (Intent To Treat Population, ITT) were included in the efficacy analyses. Participants with missing Mayo score were defined as not having achieved clinical response, remission, or mucosal healing.
Measure: Number; unit: participants
Groups:
- Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). Following this, on Days IP-29 and IP-57 abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 140 | 137 | 69 | 139
participants | 30 | 26 | 14 | 41
Statistical Analysis 1: Comparison: Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg vs IP1C-Placebo; Null hypothesis=no treatment difference between ABA arm and placebo (PLA) arm. ABA 30/~10 mg/kg vs PLA: power=98%, sample size=140 per arm,expected PLA response rate=40%, ABA 30/~10 mg/kg=65%. ABA ~10 mg/kg vs. PLA: power=90%, sample size=140 per arm, 5% significance; expected PLA response rate= 40%, ABA ~10=60%; Test type: Superiority or Other; p = 0.124, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel Chi square p-value and RR along with 95% confidence interval provided, adjusting for randomization strata (whether a participant had an inadequate response and/or intolerance to anti-TNF therapy); Conditional on ABA 30/~10 mg/kg vs PLA comparison being statistically significant at 5% level, ABA ~10 vs PLA to be tested at 5% significance level; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.48 to 1.09]

2. Secondary Outcome: IP; Baseline Mayo Score: IP1C
Description: as for outcome 1
Time Frame: Baseline
Population: The As Treated analysis population was used for all safety summaries and was defined to include all participants who received at least one infusion of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IP1C-ABA 30/~10 mg/kg: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). Following this, on Days IP-29 and IP-57 abatacept was administered IV at a dose of ~10 mg/kg.
- IP1C-ABA ~10 mg/kg: During IP, abatacept was administered IV on Days IP-1 and IP-15 at a dose of ~10 mg/kg (weight-tiered). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
- IP1C-ABA 3 mg/kg,: During IP, abatacept was administered IV on Days IP-1 and IP-15 at a dose of 3 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of 3 mg/kg.
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo
Number analyzed (Participants) | 141 | 139 | 70 | 140
units on a scale | 8.9 (1.74) | 8.8 (1.73) | 8.6 (1.82) | 8.8 (1.59)

3. Secondary Outcome: IP; Number of Participants in Clinical Remission (Per Mayo Score) at Week 12: IP1C
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. Clinical remission is defined as a Mayo score of ≤ 2 points with no individual subscore exceeding 1 point.
Time Frame: Week 12 (Day IP-85)
Population: All participants in the ITT Population were included in the efficacy analyses. Participants with missing Mayo score were defined as not having achieved clinical response, remission, or mucosal healing.
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 140 | 137 | 69 | 139
participants | 3 | 6 | 4 | 15
Statistical Analysis 1: Comparison: Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg vs IP1C-Placebo; Null hypothesis=no treatment difference between each of the ABA and placebo (PLA). At 5% significance level, Aba 30/~10 vs. PLA: power=96%, sample size=140 per arm, expected PLA rate=15%. ABA 30/~10 =35%; Aba ~10 vs. PLA: power=82%, sample size=140 per arm, expected PLA response rate= 15%, ABA/~10 mg/kg=30%; Test type: Superiority or Other; Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel Chi square p-value and RR along with 95% confidence interval provided, adjusting for randomization strata; Conditional on ABA 30/~10 vs PLA comparison for clinical response being significant at 5% level, this comparison for remission will be tested at 5%; Risk Ratio (RR) = 0.2, 95% CI 2-sided [.06 to 0.67] — Conditional on both the remission comparison for ABA 30/~10 vs PLA, and the clinical response comparison for ABA~10 vs PLA being significant at 5%, the secondary remission comparison for ABA ~10 vs PLA will be tested at 5%

4. Secondary Outcome: IP; Number of Participants in Mucosal Healing (Per Mayo Score) at Week 12: IP1C
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. Mucosal healing was defined as endoscopic subscore ≤ 1 point
Time Frame: Week 12 (Day IP-85)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 140 | 137 | 69 | 139
participants | 24 | 20 | 11 | 36
Statistical Analysis 1: Comparison: Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg vs IP1C-Placebo; Null hypothesis=no treatment difference (relative risk [RR] of ABA over placebo=1) for mucosal healing. ABA 30/~10 vs. placebo: power=99%, sample size=140 per arm, expected PLA response rate=30%, ABA 30/~10 mg/kg=60%. ABA ~10 vs. placebo: power=98%, sample size=140 per arm, 5% significance; expected PLA response rate= 30%, ABA ~10 mg/kg=55%; Test type: Superiority or Other; Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; If ABA 30/~10 vs PLA remission comparison is significant at 5% level, the mucosal healing comparison for the same treatment group will be tested at 5%; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.42 to 1.05] — Conditional on both the comparison for mucosal healing for ABA 30/~10 vs PLA and the comparison for remission for ABA ~10 vs. PLA being significant, the comparison for mucosal healing for ABA ~10 vs PLA will be tested at 5%

5. Secondary Outcome: IP; Number of Participants With Clinical Response (Per Mayo Score) at Week 12 Analyzed by Cochran-Armitage Trend Test for Dose-Response Relationship: IP1C
Description: as for outcome 1
Time Frame: Week 12 (Day IP-85)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- IP1C-ABA 3 mg/kg: During IP, abatacept was administered IV on Days IP-1 and IP-15 at a dose of 3 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of 3 mg/kg.
Arm/Group | IP1C-Placebo | IP1C-ABA 3 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 30/~10 mg/kg
Number analyzed (Participants) | 139 | 69 | 137 | 140
participants | 41 | 14 | 26 | 30
Statistical Analysis 1: Comparison: IP1C-Placebo vs IP1C-ABA 3 mg/kg vs IP1C-ABA ~10 mg/kg vs IP1C-ABA 30/~10 mg/kg; The Cochran-Armitage trend test was performed to evaluate whether a relationship existed between the response and dose regimen by comparing the proportion of participants in response across all four treatment arms; Test type: Superiority or Other; p = 0.044, Cochran-Armitage Trend Test — All statistical testing was performed at a pre-specified alpha-level of 5%

6. Secondary Outcome: IP; Baseline Inflammatory Bowel Disease Questionnaire (IBDQ) Score: IP1C
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) was used to measure disease specific quality of life. The IBDQ consists of a self-administered 32-item questionnaire that evaluates quality of life across 4 dimensional scores: Bowel, Systemic, Social and Emotional. The response to each question can range from 1 to 7, with 1 indicating severe problem and 7 indicating normal health. The total IBDQ is computed as the sum of the responses to the individual IBDQ questions. The total score can range between 32 to 224 with higher scores indicating a better quality of life.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo
Number analyzed (Participants) | 141 | 139 | 70 | 140
units on a scale | 120.0 (35.43) | 121.5 (36.42) | 126.9 (35.93) | 124.3 (33.43)

7. Secondary Outcome: IP; Mean Change From Baseline To Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ): IP1C
Description: as for outcome 6
Time Frame: Baseline (Day IP-1), Day IP-85 (Week 12)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 97 | 99 | 46 | 112
units on a scale | 9.45 (3.514) | 13.36 (3.476) | 9.87 (5.108) | 23.68 (3.268)

8. Secondary Outcome: IP; Number of Participants With Mayo Rectal Bleeding Subscores Indicating Mild Disease (≤1 Point) at Week 12: IP1C
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. An absolute rectal bleeding subscore of ≤1 point was indicative of mild disease.
Time Frame: Day IP-85 (Week 12)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 104 | 106 | 53 | 118
participants
  Rectal Subscore=0 | 28 | 36 | 16 | 47
  Rectal Subscore=1 | 31 | 30 | 13 | 27

9. Secondary Outcome: IP; Number of Participants With Mayo Stool Frequency Subscores Indicating Mild Disease (≤1 Point) at Week 12: IP1C
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. An absolute stool frequency subscore of ≤1 point was indicative of mild disease.
Time Frame: Day IP-85 (Week 12)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 104 | 106 | 53 | 118
participants
  Stool Frequency Subscore=0 | 13 | 8 | 4 | 14
  Stool Frequency Subscore=1 | 14 | 21 | 10 | 32

10. Secondary Outcome: IP; Number of Participants With Mayo Physician Global Assessment (PGA) Subscores Indicating Mild Disease (≤1 Point) at Week 12: IP1C
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. An absolute PGA subscore of ≤1 point was indicative of mild disease.
Time Frame: Day IP-85 (Week 12)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 104 | 106 | 53 | 118
participants
  PGA Subscore=0 | 2 | 4 | 3 | 11
  PGA Subscore=1 | 22 | 25 | 15 | 34

11. Secondary Outcome: IP; Number of Participants Who Are Anti-TNF-Inadequate Responders/Anti-TNF Intolerant With Clinical Response At Week 12 Analyzed by Cochran-Armitage Trend Test for Dose-Response Relationship: IP1C
Description: The Mayo Scoring system (range 0-12 points, high scores=greater severity of disease) is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Clinical response=reduction from baseline in the Mayo score of ≥ 3 points and ≥ 30%, with accompanying decrease in the rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point. Inadequate response/intolerance=inadequate response/intolerance to an approved anti-TNF agent prior to this study at an approved labeled dose for ≥8 weeks.
Time Frame: Week 12 (Day IP-85)
Population: All participants in ITT Population were included in the efficacy analyses. Participants with missing Mayo score were defined as not having achieved clinical response, remission, or mucosal healing. Prior inadequate response/intolerance was to an approved anti-TNF agent at an approved labeled dose for ≥8 weeks.
Measure: Number; unit: participants
Arm/Group | IP1C-Placebo | IP1C-ABA 3 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 30/~10 mg/kg
Number analyzed (Participants) | 45 | 24 | 46 | 45
participants | 12 | 4 | 7 | 8
Statistical Analysis 1: Comparison: IP1C-Placebo vs IP1C-ABA 3 mg/kg vs IP1C-ABA ~10 mg/kg vs IP1C-ABA 30/~10 mg/kg; The Cochran-Armitage trend test was performed to evaluate whether a relationship existed between the response and dose regimen by comparing the proportion of participants in response across all four treatment arms. Normal approximation was used if the number of responses in a treatment group is at least 5. Otherwise an exact method was used; Test type: Superiority or Other; p = 0.149, Cochran-Armitage Trend Test — All statistical testing was performed at a pre-specified alpha-level of 5%

12. Secondary Outcome: IP; Number of Participants With Clinical Response At Week 12 Among Participants With Anti-TNF (Infliximab) Failure/Intolerance: IP1C
Description: as for outcome 11
Time Frame: Week 12 (Day IP-85)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 45 | 46 | 24 | 45
participants | 8 | 7 | 4 | 12

13. Primary Outcome: Maintenance Period (MP); Number of Participants With Clinical Response (Per Mayo Score) at Month 12
Description: as for outcome 1
Time Frame: Month 12 (Day MP-365)
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- ABA ~10 mg/kg, MP: During MP, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered) every 28 days beginning Day MP-1.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 64 | 64
participants | 11 | 11

14. Secondary Outcome: IP; Number of Participants in Clinical Remission at Week 12 Among Participants With Anti-TNF (Infliximab) Failure/Intolerance: IP1C
Description: The Mayo Scoring system (range 0-12 points, high scores=greater severity of disease) is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Clinical remission is defined as a Mayo score of ≤ 2 points with no individual subscore exceeding 1 point. Inadequate response/intolerance
  =inadequate response/intolerance to an approved anti-TNF agent prior to this study at an approved labeled dose for ≥8 weeks.
Time Frame: Week 12 (Day IP-85)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 45 | 46 | 24 | 45
participants | 2 | 0 | 0 | 4

15. Primary Outcome: Open-Label Extension Period (OL); Number of Participants With Adverse Events (AEs), Related AEs, Deaths, Serious AEs (SAEs), Related SAEs, and AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: Day OL-1 through the end of the OL
Population: All participants who received at least 1 infusion of open-label study medication at any time were included in the safety analyses of the Open-Label Extension phase.
Measure: Number; unit: participants
Groups:
- ABA ~10 mg/kg, OL: During OL, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered) every 28 days beginning Day OL-1.
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 349
participants
  AEs | 241
  Related AEs | 100
  Deaths | 1
  SAEs | 66
  Related SAEs | 9
  AEs Leading to Discontinuation | 7
  SAEs Leading to Discontinuation | 4

16. Primary Outcome: OL; Number of Participants With AEs of Special Interest
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including all infections, serious infections, and opportunistic infections; autoimmune disorders; neoplasms; acute infusional AEs (pre-specified AEs occurring within 1 hour of start of infusion) and peri-infusional AEs (pre-specified AEs occurring within 24 hours of the start of infusion).
Time Frame: Day OL-1 through Day OL-729
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 349
participants
  Infections and Infestations | 127
  Serious Infections | 9
  Opportunistic Infections-Total | 2
  Opportunistic Infections-cytomegalovirus | 1
  Opportunistic Infections-listeriosis | 1
  Malignancies-Total | 5
  Malignancies-Basal Cell Carcinoma | 2
  Malignancies-Bowen's Disease | 1
  Malignancies-Chronic Myeloid Leukemia | 1
  Malignancies-Squamous Cell Carcinoma | 1
  Autoimmune Disorders-Total | 5
  Autoimmune Disorders-episcleritis | 2
  Autoimmune Disorders-scleritis | 1
  Autoimmune Disorders-anemia hemolytic autoimmune | 1
  Autoimmune Disorders-psoriasis | 1
  Acute Infusional AEs | 12
  Peri-infusional AEs | 25

17. Secondary Outcome: IP; Number of Participants in Mucosal Healing at Week 12 Among Participants With Anti-TNF (Infliximab) Failure/Intolerance: IP1C
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. Mucosal healing was defined as endoscopic subscore ≤ 1 point. Inadequate response/intolerance = inadequate response/intolerance to an approved anti-TNF agent prior to this study at an approved labeled dose for ≥8 weeks.
Time Frame: Week 12 (Day IP-85)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Induction Period Cohort 1 (IP1C)-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg | IP1C-Placebo
Number analyzed (Participants) | 45 | 46 | 24 | 45
participants | 4 | 4 | 1 | 13

18. Secondary Outcome: IP; Number of Participants With Adverse Events (AEs), Related AEs, Deaths, Serious AEs (SAEs), Related SAEs, and AEs Leading to Discontinuation: IP1C + IP2C
Description: as for outcome 15
Time Frame: Day IP-1 through Day IP-85
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- IP2C-ABA ~10 mg/kg: During IP, abatacept was administered IV on Days IP-1 and IP-15 at a dose of ~10 mg/kg (weight-tiered). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo | IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg
Number analyzed (Participants) | 141 | 139 | 70 | 140 | 51 | 50
participants
  AEs | 85 | 92 | 39 | 86 | 26 | 27
  Related AEs | 48 | 46 | 23 | 37 | 10 | 11
  Deaths | 1 | 0 | 0 | 0 | 0 | 0
  SAEs | 22 | 20 | 8 | 7 | 6 | 4
  Related SAEs | 4 | 1 | 1 | 3 | 1 | 0
  AEs Leading to Discontinuation | 4 | 6 | 2 | 5 | 1 | 0
  SAEs Leading to Discontinuation | 1 | 2 | 1 | 3 | 1 | 0

19. Secondary Outcome: IP; Number of Participants With AEs Of Special Interest: IP1C + IP2C
Description: as for outcome 16
Time Frame: Day IP-1 through Day IP-85
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo | IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg
Number analyzed (Participants) | 141 | 139 | 70 | 140 | 51 | 50
participants
  Infections and Infestations | 23 | 29 | 8 | 25 | 12 | 7
  Serious Infections | 5 | 0 | 1 | 0 | 0 | 0
  Opportunistic Infections-Total | 0 | 1 | 1 | 0 | 0 | 0
  Opportunistic Infections-candidiasis | 0 | 0 | 1 | 0 | 0 | 0
  Opportunistic Infections-esophageal candidiasis | 0 | 1 | 0 | 0 | 0 | 0
  Malignancies-Total | 1 | 0 | 0 | 1 | 0 | 0
  Malignancies-basal cell carcinoma | 1 | 0 | 0 | 0 | 0 | 0
  Malignancies-malignant melanoma | 0 | 0 | 0 | 1 | 0 | 0
  Autoimmune Disorders-Total | 2 | 1 | 0 | 4 | 0 | 0
  Autoimmune Disorders-uveitis | 1 | 1 | 0 | 1 | 0 | 0
  Autoimmune Disorders-episcleritis | 0 | 0 | 0 | 1 | 0 | 0
  Autoimmune Disorders-scleritis | 0 | 0 | 0 | 1 | 0 | 0
  Autoimmune Disorders-rheumatoid arthritis | 0 | 0 | 0 | 1 | 0 | 0
  Autoimmune Disorders-psoriasis | 1 | 0 | 0 | 0 | 0 | 0
  Acute Infusional AEs | 4 | 4 | 0 | 2 | 0 | 0
  Peri Infusional AEs | 17 | 20 | 5 | 14 | 2 | 4

20. Secondary Outcome: IP; Number of Participants With Physical Examination Findings: IP1C + IP2C
Description: Complete physical examination was obtained at the Screening Visit, Day MP-365, and OL Final Visit/Early Termination visits. Interim physical examinations were performed at other study visits. Interim physical exam were not as comprehensive as the initial full examination but did note any changes in the participant's condition since the last assessment and did not preclude examination of any of the body systems as clinically indicated. Participants were observed for AEs and vital signs (blood pressure, heart rate, and temperature).
Time Frame: Day IP-1 through Day IP-85
Population: As the results of this study were presented in a synoptic report, physical examination evaluations were not summarized. Laboratory abnormalities and vital signs were collected and summarized.
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo | IP Cohort 2 (IP2C)-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: IP; Number of Participants With Marked Hematology Laboratory Abnormalities: IP1C
Description: High=greater than Upper Normal Limit (ULN), Low=lower than Lower Normal Limit (LLN). LLN/ULN= Hemoglobin (HGB): >3 g/dL decrease from Baseline (BL); Hematocrit: <0.75 x BL; Erythrocytes: <0.75 x BL; Platelets (PLT): <0.67 x LLN/>1.5 x ULN; Leukocytes: <0.75 x LLN/ >1.25 x ULN; neutrophils+bands: <1.0 x 10^3 c/uL; eosinophils: >0.750 x 10^3 c/uL; monocytes: >2000 mm3; lymphocytes: <0.750 x 10^3 c/uL/ >7.50 x 10^3 c/uL.
Time Frame: Day IP-1 through Day IP-85
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo
Number analyzed (Participants) | 141 | 139 | 70 | 140
participants
  Low HGB; n=136, n=134, n=67, n=133 | 3 | 2 | 6 | 1
  Low hematocrit; n=134, n=133, n=67, n=131 | 1 | 2 | 4 | 1
  Low erythrocytes; n=136, n=134, n=67, n=133 | 2 | 2 | 4 | 1
  Low PLT; n=136, n=133, n=66, n=133 | 1 | 0 | 1 | 0
  High PLT; n=136, n=133, n=66, n=133 | 0 | 2 | 0 | 0
  Low leukocytes; n=136, n=134, n=67, n=133 | 1 | 0 | 4 | 1
  High leukocytes; n=136, n=134, n=67, n=133 | 10 | 6 | 3 | 5
  Low neutrophils + bands; n=136, n=134, n=67, n=131 | 0 | 0 | 1 | 0
  High eosinophils; n=136, n=134, n=67, n=131 | 6 | 4 | 3 | 4
  High monocytes; n=136, n=134, n=67, n=131 | 0 | 0 | 1 | 0
  Low lymphocytes; n=136, n=134, n=67, n=131 | 23 | 13 | 11 | 26

22. Secondary Outcome: IP; Number of Participants With Marked Liver and Kidney Function and Electrolyte Laboratory Abnormalities: IP1C
Description: Low=lower than LLN, High=greater than ULN. LLN/ULN= Alkaline phosphatase (ALP): >2 x ULN; aspartate aminotransferase (AST): >3 x ULN; alanine aminotransferase (ALT): >3 x ULN; G-Glutamyl transferase (GGT): >2 x ULN; Bilirubin: >2 x ULN; blood urea nitrogen (BUN): >2 x BL; creatinine: >4 x BL; Sodium (Na): <0.95 x LLN/ >1.05 x ULN; potassium (K): <0.9 x LLN/ >1.1 x ULN; calcium (Ca): <0.8 x LLN/>1.2 x ULN; phosphorous (P): <0.75 x LLN/ >1.2 5 x ULN
Time Frame: Day IP-1 through Day IP-85
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo
Number analyzed (Participants) | 141 | 139 | 70 | 140
participants
  High ALP, n=137, n=135, n=66, n=135 | 1 | 0 | 0 | 0
  High ALT; n=137, n=135, n=66, n=135 | 0 | 1 | 0 | 0
  High GGT; n=137, n=135, n=66, n=135 | 6 | 2 | 0 | 2
  High BUN; n=127, n=130, n=62, n=124 | 0 | 2 | 2 | 3
  High creatinine; n=137, n=135, n=66, n=135 | 0 | 0 | 0 | 1
  Low Na; n=138, n=135, n=66, n=135 | 0 | 0 | 2 | 0
  Low K; n=138, n=135, n=66, n=135 | 1 | 2 | 2 | 0
  High K; n=138, n=135, n=66, n=135 | 0 | 1 | 0 | 1
  Low Ca; n=137, n=135, n=66, n=135 | 0 | 1 | 2 | 0
  Low P; n=137, 135, n=66, n=135 | 0 | 1 | 0 | 3

23. Secondary Outcome: IP; Number of Participants With Marked Chemistry and Urinalysis Laboratory Abnormalities: IP1C
Description: Low=lower than LLN, High=greater than ULN. LLN/ULN= serum glucose (Glu): <65 mg/dL/ >220 mg/dL; total protein: < 0.9 x LLN/ >1.1 x ULN; albumin:<0.9 x LLN; uric acid: >1.5 x ULN. For Urinalysis (Urine protein, urine Glu, urine blood, leukocyte esterase, Red Blood Cells [RBCs], White Blood Cells [WBCs]): Use ≥2 when BL value missing or value ≥4, or when pre-dose=0 or 0.5. Use ≥3 when pre-dose=1. Use ≥4 when pre-dose=2 or 3
Time Frame: Day IP-1 through Day IP-85
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | IP1C-ABA 30/~10 mg/kg | IP1C-ABA ~10 mg/kg | IP1C-ABA 3 mg/kg, | IP1C-Placebo
Number analyzed (Participants) | 141 | 139 | 70 | 140
participants
  Low Glu; n=88, n=91, n=41, n=105 | 1 | 6 | 2 | 0
  High Glu; n=88, n=91, n=41, n=105 | 0 | 0 | 1 | 0
  Low protein; n=137, n=135, n=66, n=135 | 5 | 3 | 3 | 0
  High protein; n=137, n=135, n=66, n=135 | 0 | 1 | 0 | 0
  Low albumin; n=137, n=135, n=66, n=135 | 7 | 5 | 3 | 0
  High urine protein; n=132, n=129, n=66, n=128 | 5 | 3 | 2 | 4
  High urine Glu; n=132, n=129, n=66, n=128 | 4 | 1 | 2 | 4
  High urine blood; n=132, n=129, n=66, n=128 | 6 | 7 | 4 | 11
  High leukocyte esterase; n=54, n=51, n=27, n=52 | 1 | 5 | 2 | 2
  High urine RBC; n=47, n=42, n=17, n=52 | 9 | 8 | 4 | 12
  High urine WBC; n=64, n=56, n=27, n=58 | 14 | 21 | 3 | 14

24. Secondary Outcome: IP; Number of Participants With Marked Hematology, Liver and Kidney Function, and Electrolyte Laboratory Abnormalities: IP2C
Description: High=greater than Upper Normal Limit (ULN), Low=lower than Lower Normal Limit (LLN). LLN/ULN= Hemoglobin (HGB): >3 g/dL decrease from Baseline (BL); Hematocrit: <0.75 x BL; Erythrocytes: <0.75 x BL; Platelets (PLT): <0.67 x LLN/>1.5 x ULN; Leukocytes: <0.75 x LLN/ >1.25 x ULN; eosinophils: >0.750 x 10^3 c/uL; monocytes: >2000 mm3; lymphocytes: <0.750 x 10^3 c/uL/ >7.50 x 10^3 c/uL; blood urea nitrogen (BUN): >2 x BL; creatinine: >4 x BL; Sodium (Na): <0.95 x LLN/ >1.05 x ULN; potassium (K): <0.9 x LLN/ >1.1 x ULN; phosphorous (P): <0.75 x LLN/ >1.2 5 x ULN;
Time Frame: Day IP-1 through Day IP-85
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- IP2C-ABA 30/~10 mg/kg: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). Following this, on Days IP-29 and IP-57 abatacept was administered IV at a dose of ~10 mg/kg.
Arm/Group | IP2C-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg
Number analyzed (Participants) | 51 | 50
participants
  Low HGB; n=50, n=49 | 2 | 2
  Low hematocrit; n=50, n=49 | 1 | 0
  Low erythrocytes; n=50, n=49 | 1 | 0
  High PLT; n=50, n=49 | 0 | 1
  Low leukocytes; n=50, n=49 | 0 | 1
  High leukocytes; n=50, n=49 | 3 | 4
  High eosinophils; n=49, n=49 | 3 | 1
  High monocytes; n=49, n=49 | 0 | 1
  Low lymphocytes; n=49, n=49 | 5 | 3
  High BUN; n=46, n=44 | 3 | 1
  High creatinine; n=50, n=50 | 1 | 0
  Low Na; n=50, n=50 | 1 | 0
  Low K; n=50, n=50 | 2 | 1
  Low P; n=50, n=50 | 1 | 0
  Low Glu; n=37, n=28 | 0 | 2
  High Glu; n=37, n=28 | 0 | 2
  Low protein; n=50, n=50 | 2 | 0
  Low albumin; n=50, n=50 | 2 | 0
  High urine protein; n=50, n=48 | 0 | 4
  High urine Glu; n=50, n=48 | 0 | 2
  High urine blood; n=50, n=48 | 2 | 3
  High leukocyte esterase; n=21, n=16 | 4 | 2
  High urine RBC; n=15, n=20 | 0 | 4
  High urine WBC; n=24, n=23 | 7 | 6

25. Secondary Outcome: IP; Number of Participants With Marked Chemistry and Urinalysis Laboratory Abnormalities: IP2C
Description: Low=lower than LLN, High=greater than ULN. LLN/ULN= serum glucose (Glu): <65 mg/dL/ >220 mg/dL; total protein: < 0.9 x LLN/ >1.1 x ULN; albumin:<0.9 x LLN. For Urinalysis (Urine protein, urine Glu, urine blood, leukocyte esterase, Red Blood Cells [RBCs], White Blood Cells [WBCs]): Use ≥2 when BL value missing or value ≥4, or when pre-dose=0 or 0.5. Use ≥3 when pre-dose=1. Use ≥4 when pre-dose=2 or 3
Time Frame: Day IP-1 through Day IP-85
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | IP2C-ABA 30/~10 mg/kg | IP2C-ABA ~10 mg/kg
Number analyzed (Participants) | 51 | 50
participants
  Low Glu; n=37, n=28 | 0 | 2
  High Glu; n=37, n=28 | 0 | 2
  Low protein; n=50, n=50 | 2 | 0
  Low albumin; n=50, n=50 | 2 | 0
  High urine protein; n=50, n=48 | 0 | 4
  High urine Glu; n=50, n=48 | 0 | 2
  High urine blood; n=50, n=48 | 2 | 3
  High leukocyte esterase; n=21, n=16 | 4 | 2
  High urine RBC; n=15, n=20 | 0 | 4
  High urine WBC; n=24, n=23 | 7 | 6

26. Secondary Outcome: IP; Number of Participants With Abatacept-Induced Antibodies: IP1C + IP2C
Description: A electrochemiluminescent immunoassay screened sera for drug-specific antibodies, immunocompetition was used to identify specific anti-Abatacept reactivity. CTLA4 and Possibly Ig category=reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; Abatacept molecule). Ig and/or Junction category=reactivity against constant regions and/or hinge region of human IgG1. Drug-induced seropositivity was defined as a post-baseline titer higher than Baseline, or any post-baseline positivity if Baseline value was missing.
Time Frame: For participants treated in MP: Day IP-1 (Baseline) to Day MP-1 (Day IP-85). For participants treated in OL directly after IP: Day IP-1 to Day OL-1. For participants treated only in IP: All measurements after Day IP-1 (including follow-up visits)
Population: All subjects with at least one post-baseline immunogenicity measurement during the study period were included in the immunogenicity data set. "Positive" was defined as "positive post-baseline IP-1" and with a titer value greater than the baseline titer value. Participants with missing baseline titer were assumed "negative" at baseline.
Measure: Number; unit: participants
Groups:
- IP1C+IP2C: ABA 30/~10 mg/kg: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). Following this, on Days IP-29 and IP-57 abatacept was administered IV at a dose of ~10 mg/kg.
- IP1C+IP2C: ABA ~10 mg/kg: During IP, abatacept was administered IV on Days IP-1 and IP-15 at a dose of ~10 mg/kg (weight-tiered). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
Arm/Group | IP1C+IP2C: ABA 30/~10 mg/kg | IP1C+IP2C: ABA ~10 mg/kg | IP1C-ABA 3 mg/kg
Number analyzed (Participants) | 189 | 185 | 66
participants
  Total | 6 | 19 | 4
  CTLA4/Possibly Ig | 2 | 17 | 4
  Ig and/or Ig Junction | 4 | 3 | 0

27. Secondary Outcome: MP; Number of Participants in Clinical Remission at Month 12
Description: as for outcome 3
Time Frame: Month 12 (Day MP-365)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 64 | 64
participants | 8 | 9

28. Secondary Outcome: MP; Number of Participants With Mayo Endoscopic Subscores Indicating Mucosal Healing (≤1 Point) at Month 12
Description: as for outcome 4
Time Frame: Month 12 (Day MP-365)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 17 | 12
participants | 11 | 10

29. Secondary Outcome: MP; Number of Participants in Clinical Remission at Both Month 6 and Month 12
Description: as for outcome 3
Time Frame: Month 6 (Day MP-169), Month 12 (Day MP-365)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis to determine the percentage of participants in clinical remission at both Month 6 and Month 12 was not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: MP; Number of Participants With Baseline Oral Corticosteroid Use Who Have Discontinued Corticosteroids and Achieved Clinical Remission by Month 12
Description: Baseline corticosteroids equivalent of ≤30 mg prednisone daily. The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater frequency or severity. Clinical remission is defined as a Mayo score of ≤ 2 points with no individual subscore exceeding 1 point.
Time Frame: Day MP-365 (Month 12)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analyses for corticosteroid sparing were not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: MP; Mean Change From Baseline to Month 12 in IBDQ
Description: as for outcome 6
Time Frame: Day MP-365
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis for changes from baseline in IBDQ responses were not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: MP; Mean Change From Baseline to Month 12 in Short Form-36 (SF-36)
Description: The SF-36 is a validated instrument to measure health-related quality of life across multiple disease states. Individual subscale scores and 2 summary scores are calculated: (1) physical component summary (PCS) which includes physical functioning, role-physical, bodily pain, and general health; (2) mental component summary (MCS) which includes vitality, social functioning, role-emotional, and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight, with values ranging from worse health (0) to best health (100).
Time Frame: Day MP-365
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis for changes from baseline in SF-36 responses were not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: MP; Number of Participants With Baseline Oral Corticosteroid Use Who Have Discontinued Corticosteroids for 90 Consecutive Days and Achieved Clinical Remission by Month 12
Description: as for outcome 30
Time Frame: Day MP-365 (Month 12)
Population: as for outcome 30
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: MP; Number of Participants With Mayo Rectal Bleeding Subscores Indicating Mild Disease (≤1 Point) at Month 12
Description: as for outcome 8
Time Frame: Day MP-365 (Month 12)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis to determine the percentage of participants with rectal subscores indicating mild disease (≤1) was not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: MP; Number of Participants With Mayo Stool Frequency Subscores Indicating Mild Disease (≤1 Point) at Month 12
Description: as for outcome 9
Time Frame: Day MP-365 (Month 12)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis to determine the percentage of participants with stool frequency subscores indicating mild disease (≤1) was not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: MP; Number of Participants With Mayo PGA Subscores Indicating Mild Disease (≤1 Point) at Month 12
Description: as for outcome 10
Time Frame: Day MP-365 (Month 12)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis to determine the percentage of participants with PGA subscores indicating mild disease (≤1) was not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: MP; Number of Participants With Clinical Response at Month 12 Among Participants With Inadequate Response/Intolerance to Prior Anti-TNF Therapy (Infliximab)
Description: as for outcome 11
Time Frame: Month 12 (Day MP-365)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary subgroup analyses of clinical response in subjects who have had an inadequate response and/or intolerance to anti-TNF therapy was not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: MP; Number of Participants With Clinical Remission at Month 12 Among Participants With Inadequate Response/Intolerance to Prior Anti-TNF Therapy (Infliximab)
Description: as for outcome 14
Time Frame: Month 12 (Day MP-365)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary subgroup analyses of clinical remission in subjects who have had an inadequate response and/or intolerance to anti-TNF therapy was not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: MP; Number of Participants With Clinical Mucosal Healing at Month 12 Among Participants With Inadequate Response/Intolerance to Prior Anti-TNF Therapy (Infliximab)
Description: The Mayo Scoring system ranges from 0 - 12 points and is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Higher Mayo scores indicate greater severity of disease. Mucosal healing was defined as endoscopic subscore ≤1 point. Inadequate response/intolerance = inadequate response/intolerance to an approved anti-TNF agent prior to this study at an approved labeled dose for ≥8 weeks.
Time Frame: Month 12 (Day MP-365)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary subgroup analyses of mucosal healing in subjects who have had an inadequate response and/or intolerance to anti-TNF therapy was not conducted for the MP as planned.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: MP; Number of Participants With Abatacept-Induced Antibodies
Description: as for outcome 26
Time Frame: For participants not entering OL: All measurements starting after Day MP-1 (including follow-up visits). For participants entering OL: From first measurement after Day MP-1 to Day MP-365 (Day OL-1).
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 62 | 47
participants
  Total | 8 | 20
  CTLA4/Possibly Ig | 8 | 17
  Ig and/or Ig Junction | 0 | 3

41. Secondary Outcome: MP; Number of Participants With Adverse Events (AEs), Related AEs, Deaths, Serious AEs (SAEs), Related SAEs, and AEs Leading to Discontinuation
Description: as for outcome 15
Time Frame: Day MP-1 through Day MP-365
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 65 | 66
participants
  AEs | 39 | 36
  Related AEs | 12 | 13
  Deaths | 1 | 0
  SAEs | 7 | 4
  Related SAEs | 2 | 2
  AEs Leading to Discontinuation | 1 | 3
  SAEs Leading to Discontinuation | 1 | 1

42. Secondary Outcome: MP; Number of Participants With AEs of Special Interest
Description: as for outcome 16
Time Frame: Day MP-1 through Day MP-365
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 65 | 66
participants
  Infections and Infestations | 39 | 36
  Serious Infections | 5 | 2
  Opportunistic Infections-Total | 1 | 0
  Opportunistic Infections-pneumonia herpes viral | 1 | 0
  Malignancies-Total | 0 | 1
  Malignancies-breast cancer | 0 | 1
  Autoimmune Disorders-Total | 2 | 0
  Autoimmune Disorders-erythema nodosum | 1 | 0
  Autoimmune Disorders-pemphigoid | 1 | 0
  Acute Infusional AEs | 2 | 1
  Peri-infusional AEs | 3 | 2

43. Secondary Outcome: MP; Number of Participants With Physical Examination Findings
Description: as for outcome 20
Time Frame: Day IP-85 through Day MP-365
Population: as for outcome 20
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: MP; Number of Participants With Marked Hematology Laboratory Abnormalities
Description: High=greater than ULN, Low=lower than LLN. LLN/ULN= HGB: >3 g/dL decrease from Baseline (BL); Hematocrit: <0.75 x BL; Erythrocytes: <0.75 x BL; PLT: <0.67 x LLN/>1.5 x ULN; Leukocytes: <0.75 x LLN/ >1.25 x ULN; neutrophils+bands: <1.0 x 10^3 c/uL; eosinophils: >0.750 x 10^3 c/uL; monocytes: >2000 mm3; lymphocytes: <0.750 x 10^3 c/uL/ >7.50 x 10^3 c/uL; GGT: >2 x ULN; Bilirubin: >2 x ULN; BUN: >2 x BL; Na: <0.95 x LLN/ >1.05 x ULN; K: <0.9 x LLN/ >1.1 x ULN; Ca: <0.8 x LLN/>1.2 x ULN
Time Frame: Day IP-85 through Day MP-365
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- ABA 30/~10 mg/kg, MP: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). Following this, on Days IP-29 and IP-57 abatacept was administered IV at a dose of ~10 mg/kg.
- ABA ~10 mg/kg, MP: During IP, abatacept was administered IV on Days IP-1 and IP-15 at a dose of ~10 mg/kg (weight-tiered). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
Arm/Group | ABA 30/~10 mg/kg, MP | ABA ~10 mg/kg, MP
Number analyzed (Participants) | 65 | 66
participants
  Low HGB; n=64, n=61 | 1 | 2
  Low hematocrit; n=64, n=60 | 3 | 2
  Low erythrocytes; n=64, n=61 | 1 | 2
  High PLT; n= 64, n=61 | 0 | 1
  Low leukocytes; n=64, n=60 | 2 | 0
  High leukocytes; n=64, n=60 | 2 | 0
  Low neutrophils + bands; n=64, n=60 | 1 | 0
  High eosinophils; n=64, n=60 | 2 | 3
  High monocytes; n=64, n=60 | 1 | 0
  Low lymphocytes; n=64, n=60 | 7 | 6
  High lymphocytes; n=64, n=60 | 1 | 0
  High GGT; n=64, n=62 | 3 | 2
  High bilirubin, n=64, n=61 | 1 | 0
  High BUN; n=57, n=59 | 4 | 3
  Low Na; n=64, n=62 | 0 | 1
  Low K; n=64, n=62 | 1 | 1
  Low Ca; n=64, n=61 | 1 | 0
  Low Glu; n=45, n=38 | 0 | 2
  High Glu; n=45, n=38 | 3 | 3
  Low protein; n=64, n=61 | 0 | 1
  High urine protein; n=58, n=58 | 4 | 1
  High urine Glu; n=58, n=58 | 2 | 1
  High urine blood; n=58, n=58 | 3 | 7
  High leukocyte esterase; n=23, n=18 | 2 | 5
  High urine RBC; n=24, n=17 | 4 | 4
  High urine WBC; n=29, n=21 | 8 | 10

45. Secondary Outcome: MP; Number of Participants With Marked Chemistry and Urinalysis Laboratory Abnormalities
Description: Low=lower than LLN, High=greater than ULN. LLN/ULN= serum glucose (Glu): <65 mg/dL/ >220 mg/dL; fasting serum Glu: <0.8 x LLN/ >1.5 x ULN; total protein: < 0.9 x LLN/ >1.1 x ULN; albumin:<0.9 x LLN; uric acid: >1.5 x ULN. For Urinalysis (Urine protein, urine Glu, urine blood, leukocyte esterase, Red Blood Cells [RBCs], White Blood Cells [WBCs]): Use ≥2 when BL value missing or value ≥4, or when pre-dose=0 or 0.5. Use ≥3 when pre-dose=1. Use ≥4 when pre-dose=2 or 3
Time Frame: Day IP-85 through Day MP-365
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | ABA 30/~10 mg/kg, MP | ABA ~10 mg/kg, MP
Number analyzed (Participants) | 65 | 66
participants
  Low Glu; n=45, n=38 | 0 | 2
  High Glu; n=45, n=38 | 3 | 3
  Low protein; n=64, n=61 | 0 | 1
  High urine protein; n=58, n=58 | 4 | 1
  High urine Glu; n=58, n=58 | 2 | 1
  High urine blood; n=58, n=58 | 3 | 7
  High leukocyte esterase; n=23, n=18 | 2 | 5
  High urine RBC; n=24, n=17 | 4 | 4
  High urine WBC; n=29, n=21 | 8 | 10

46. Primary Outcome: OL; Number of Participants With Physical Examination Findings
Description: as for outcome 20
Time Frame: Day OL-1 through Day OL-729
Population: as for outcome 20
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: OL; Number of Participants With Clinical Response Over Time
Description: as for outcome 1
Time Frame: Day OL-1 through Day OL-729
Population: All participants who received at least 1 infusion of open-label study medication at any time were included in the efficacy analyses of the OL. Number of Participants Analyzed=all participants in OL; n=number of evaluable participants.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 347
participants
  Day OL-365 (n=163) | 44
  Day OL-729 (n=4) | 0

48. Secondary Outcome: OL; Number of Participants With Clinical Remission Over Time
Description: as for outcome 3
Time Frame: Day OL-1 through Day OL-729
Population: as for outcome 47
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 347
participants
  Day OL-365 (n=163) | 18
  Day OL-729 (n=4) | 0

49. Primary Outcome: OL; Number of Participants With Marked Hematology Laboratory Abnormalities
Description: as for outcome 21
Time Frame: Day OL-1 through Day OL-729
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- ABA ~10 mg/kg, OL: During IP, abatacept was administered IV on Days IP-1 and IP-15 at a dose of ~10 mg/kg (weight-tiered). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 349
participants
  Low HGB; n=326 | 20
  Low hematocrit; n=322 | 17
  Low erythrocytes; n=326 | 6
  High PLT; n=323 | 3
  Low leukocytes; n=326 | 3
  High leukocytes; n=326 | 18
  Low neutrophils + bands; n=324 | 1
  High eosinophils; n=324 | 17
  High monocytes; n=324 | 2
  Low lymphocytes; n=324 | 43

50. Primary Outcome: OL; Number of Participants With Liver and Kidney Function and Electrolyte Laboratory Abnormalities
Description: Low=lower than LLN, High=greater than ULN. LLN/ULN= Alkaline phosphatase (ALP): >2 x ULN; aspartate aminotransferase (AST): >3 x ULN; alanine aminotransferase (ALT): >3 x ULN; G-Glutamyl transferase (GGT): >2 x ULN; Bilirubin: >2 x ULN; blood urea nitrogen (BUN): >2 x BL; creatinine: >4 x BL; potassium (K): <0.9 x LLN/ >1.1 x ULN; calcium (Ca): <0.8 x LLN/>1.2 x ULN; phosphorous (P): <0.75 x LLN/ >1.2 5 x ULN
Time Frame: Day OL-1 through Day OL-729
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 349
participants
  High ALP, n=331 | 4
  High AST, n=331 | 3
  High ALT; n=331 | 3
  High GGT; n=332 | 17
  High bilirubin, n=331 | 1
  High BUN; n=310 | 10
  High creatinine; n=330 | 5
  Low K; n=331 | 7
  Low Ca; n=330 | 2
  Low P; n=330 | 4
  High P, n=330 | 1

51. Primary Outcome: OL; Number of Participants With Chemistry and Urinalysis Laboratory Abnormalities
Description: as for outcome 45
Time Frame: Day OL-1 through Day OL-729
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 349
participants
  Low Glu; n=245 | 4
  High Glu; n=245 | 6
  Low protein; n=331 | 3
  Low albumin; n=331 | 12
  High urine protein; n=312 | 11
  High urine Glu; n=312 | 4
  High urine blood; n=312 | 27
  High leukocyte esterase; n=122 | 10
  High urine RBC; n=115 | 22
  High urine WBC; n=150 | 45

52. Secondary Outcome: OL; Number of Participants With Mayo Endoscopic Subscores Indicating Mucosal Healing (≤1 Point) During OL
Description: as for outcome 4
Time Frame: Open-Label Period (Day OL-1 through Day OL-729)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary subgroup analyses of mucosal healing was not conducted for the OL as planned.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 17 | 12
participants | 0 | 0

53. Secondary Outcome: OL; Number of Participants With Clinical Response or Clinical Remission Upon Retreatment With Abatacept Among Those Who Received Abatacept in the IP or MP Period
Description: The Mayo Scoring system (range 0-12 points, high scores=greater severity of disease) is a composite index consisting of 4 disease variables (stool frequency, rectal bleeding, endoscopy evaluation, and Physician's Global Assessment). Clinical response=reduction from baseline in the Mayo score of ≥ 3 points and ≥ 30%, with accompanying decrease in the rectal bleeding subscore of ≥ 1 point or absolute rectal bleeding subscore of ≤ 1 point. Clinical remission = Mayo score of ≤ 2 points with no individual subscore exceeding 1 point. Change from Baseline= post-Baseline - Baseline value.
Time Frame: Last Study Visit (Day OL-729)
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary subgroup analyses of clinical efficacy upon retreatment with abatacept among participants who received study drug during the IP or MP was not conducted for the OL as planned.
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 0

54. Secondary Outcome: OL; Number of Participants With Abatacept-Induced Antibodies
Description: as for outcome 26
Time Frame: For participants receiving OL medication, all measurements starting after Day OL-1 (including follow-up visits and at 56 and 85 days after last dose)
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 324
participants
  Total | 66
  CTLA4/Possibly Ig | 59
  Ig and/or Ig Junction | 11

55. Secondary Outcome: OL; Number of Participants Using Corticosteroids During OL
Description: Participants taking oral corticosteroids (equivalent of ≤ 30 mg prednisone daily) must have met minimum treatment duration at entry into IP and had stable dose for ≥2 weeks prior to entry into the IP.
Time Frame: Day OL-1 through Day OL-729
Population: Due to the early termination of the study after preliminary IP1C results were reviewed and the primary efficacy endpoint was not achieved, the secondary subgroup analyses of corticosteroid use was not conducted for the OL as planned.
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- ABA 30/~10 mg/kg,IP1C: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered).
- ABA 30/~10mg/kg,IP2C: During IP, abatacept was administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg.
- ABA 3 mg/kg,IP1C: During IP, abatacept was administered IV on Days IP-1, IP-15, IP-29, and IP-57 at a dose of 3 mg/kg (fixed dose).
- ABA ~10 mg/kg,IP1C; ABA ~10mg/kg,IP2C: During IP, abatacept was administered IV on Days IP-1,IP-15, IP-29, and IP-57 at a dose of ~10 mg/kg (weight-tiered).
- ABA ~10mg/kg, MP: During MP, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered) every 28 days beginning Day MP-1.
- Placebo, IP1C: During the IP, placebo was administered IV on Days IP-1, IP-15, IP-29, and IP-57.
Arm/Group | ABA 30/~10 mg/kg,IP1C | ABA 30/~10mg/kg,IP2C | ABA 3 mg/kg,IP1C | ABA ~10 mg/kg,IP1C | ABA ~10mg/kg,IP2C | ABA ~10mg/kg, MP | ABA ~10 mg/kg, OL | Placebo, IP1C | Placebo, MP
Serious Adverse Events (participants affected / at risk) | 22/141 | 6/51 | 8/70 | 20/139 | 4/50 | 7/65 | 66/349 | 7/140 | 4/66
Other Adverse Events (participants affected / at risk) | 49/141 | 13/51 | 21/70 | 48/139 | 13/50 | 20/65 | 137/349 | 45/140 | 24/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABA 30/~10 mg/kg,IP1C (N=141) | ABA 30/~10mg/kg,IP2C (N=51) | ABA 3 mg/kg,IP1C (N=70) | ABA ~10 mg/kg,IP1C (N=139) | ABA ~10mg/kg,IP2C (N=50) | ABA ~10mg/kg, MP (N=65) | ABA ~10 mg/kg, OL (N=349) | Placebo, IP1C (N=140) | Placebo, MP (N=66)
VISION BLURRED (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PERSONALITY CHANGE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
PROCTALGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 13 | 5 | 5 | 14 | 4 | 3 | 42 | 4 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
VIRAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VARICELLA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LISTERIOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HIV INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PILONIDAL CYST (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PELVIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PNEUMONIA HERPES VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GLOMERULONEPHRITIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PYODERMA GANGRENOSUM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ASTHENIA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
INFUSION RELATED REACTION (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABA 30/~10 mg/kg,IP1C (N=141) | ABA 30/~10mg/kg,IP2C (N=51) | ABA 3 mg/kg,IP1C (N=70) | ABA ~10 mg/kg,IP1C (N=139) | ABA ~10mg/kg,IP2C (N=50) | ABA ~10mg/kg, MP (N=65) | ABA ~10 mg/kg, OL (N=349) | Placebo, IP1C (N=140) | Placebo, MP (N=66)
HEADACHE (Nervous system disorders) | 17 | 3 | 7 | 12 | 6 | 3 | 24 | 12 | 5
DIZZINESS (Nervous system disorders) | 4 | 1 | 4 | 2 | 0 | 0 | 7 | 3 | 3
NAUSEA (Gastrointestinal disorders) | 8 | 1 | 3 | 11 | 3 | 2 | 18 | 9 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 | 2 | 1 | 1 | 3 | 3 | 16 | 5 | 4
INFLUENZA (Infections and infestations) | 1 | 1 | 0 | 3 | 0 | 4 | 12 | 3 | 1
NASOPHARYNGITIS (Infections and infestations) | 5 | 2 | 2 | 3 | 1 | 3 | 29 | 8 | 3
URINARY TRACT INFECTION (Infections and infestations) | 5 | 2 | 3 | 4 | 3 | 0 | 11 | 1 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 1 | 2 | 0 | 2 | 22 | 5 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 0 | 4 | 13 | 3 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 6 | 0 | 2 | 18 | 4 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2 | 4 | 1 | 4 | 13 | 3 | 5
FATIGUE (General disorders) | 6 | 3 | 3 | 8 | 3 | 1 | 16 | 3 | 2
PYREXIA (General disorders) | 9 | 3 | 6 | 6 | 1 | 2 | 17 | 2 | 1
ASTHENIA (General disorders) | 8 | 0 | 1 | 4 | 0 | 0 | 6 | 2 | 1

LIMITATIONS AND CAVEATS:
This study was terminated after review of the IP1C results due to lack of efficacy. Enrollment for the MP and for IP2C was not completed. Participants in MP, IP2C, and OL were early terminated at the time of study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.